CLINICAL TRIAL: NCT06133907
Title: Investigation of the Frequency of Hereditary Hyper Alpha-tryptasemia in Patients With Elevated Basal Tryptasemia (Protocol HaT)
Brief Title: Investigation of the Frequency of Hereditary Hyper Alpha-tryptasemia in Patients With Elevated Basal Tryptasemia
Acronym: HaT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-AOI-12
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Allergic Bronchiolitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Samples Without DNA (Experimental): Patients who came to the pneumoallergology department of the CHU de Nice since January 2014 for an allergological workup and with tryptasemia was ≥ 8ng/ml (at least once in patient history).
  Interventions: Genetic: Serum

INTERVENTIONS:
Genetic: Serum — Patients who came to the pneumoallergology department of the CHU de Nice since January 2014 for an allergological workup and with tryptasemia was ≥ 8ng/ml (at least once in patient history).

SUMMARY:
The aim of the study is to assess the number of patients with elevated blood tryptase for whom this elevation could be linked to a hereditary alpha-tryptase secretion abnormality or hyper-alpha-tryptasemia. This information will enable to better optimize the management and follow-up of patients who have experienced hypersensitivity reactions and have elevated basal blood tryptase levels. The patients will be offered the opportunity to take part in the study. If they consent to participate, they will be tested for hereditary hyper-alpha-tryptasemia. A blood sampling will be performed in the center. A few weeks after, the patient will be informed about the blood sample result during a medical consultation organized in the center.

ELIGIBILITY:
Inclusion Criteria:

* Patients who came in the pneumoallergology department of the CHU de Nice since January 2014 for an allergological workup
* Patients who have received at least one basal tryptase assay, according to recommendations
* informed consent signature

Exclusion Criteria:

* High tryptasemia (≥ 8ng/ml) synchronous with anaphylactic reaction and unconfirmed basally
* Known diagnosis of systemic mastocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hereditary hyper alpha-tryptasemia | at inclusion
  Analysis machine by PCR

SECONDARY OUTCOMES:
Phenotyping our patient cohort | at 36 months
  longitudinal follow-up of clinical symptoms according to patient subgroups in relation to mast cell pathologies.
Set up a serotheque to support scientific and medical projects in this field | At inclusion
  Biobanking

CONTACTS AND LOCATIONS:
Overall Officials: Leroy Sylvie, PhD, Principal Investigator — CHU de Nice, Service de Pneumologie
Locations (1):
- CHU de Nice - Hôpital de Pasteur, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided